CLINICAL TRIAL: NCT01639469
Title: A Telemedicine Intervention to Improve Physical Function in Patients With PD
Brief Title: Telemedicine Intervention to Improve Physical Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IIR 11-342
Record Dates: First submitted 2012-07-10; First posted 2012-07-12 (Estimated); Results first posted 2017-06-23 (Actual); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Parkinson's Disease
Keywords: Parkinson Disease; Quality of Life; Exercise Therapy
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Structured exercise (Experimental): Structured exercise instruction by smartphone
  Interventions: Behavioral: Structured exercise
- lifestyle exercise (Active Comparator): Lifestyle exercise program taught via smartphone
  Interventions: Behavioral: Lifestyle exercise

INTERVENTIONS:
Behavioral: Structured exercise — Structured exercise includes stretching, strengthening, and balance exercises.
  Arms: Structured exercise
Behavioral: Lifestyle exercise — Subjects will be taught lifestyle exercises and advised about mobility strategies
  Arms: lifestyle exercise

SUMMARY:
This project is investigating whether a one-year in-home exercise program will reduce the rate of falls and improve strength and quality of life in patients with Parkinson's disease.

DETAILED DESCRIPTION:
Background/Rationale:

Parkinson's disease (PD) is the second most common neurodegenerative disease, affecting over one million Americans. The cardinal clinical manifestations of PD are motoric, which limit functional mobility leading to difficulty working, caring for family members, managing a household, and overall decreased independence and quality of life (QOL). A wealth of growing data indicates tremendous benefits of exercise for patients with PD. Not only have exercise programs been shown to improve motor function and reduce the risk of falls, but also improve overall QOL and possibly the very course of disease pathology. However, programs that involve supervision in the home of people with PD are expensive to roll out widely, and programs that involve people with PD traveling to a central site not only result in non-compliance over time because of difficulty getting to the site, but also rule out the involvement of a large number of people with PD who simply live too far from larger centers where such programs are typically established.

Objective:

The investigators hypothesize that a one-year in-home exercise program, centered around remote, real-time instruction and supervision, will reduce the rate of falls and improve strength and QOL in patients with PD.

Methods:

The proposed study is a randomized controlled trial of a structured exercise program, evaluating effects on fall rate, physical functioning, and QOL. Community-dwelling people with PD will be randomized either to a group who receives structured and remote exercise instruction and supervision in real-time or a group who is taught a lifestyle exercise program. Subjects will be male and female Veterans with a physician diagnosis of idiopathic, typical PD, with at least 2 of 3 cardinal signs of PD, and response to dopaminergic medication. The interventions will last one year.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of idiopathic, typical Parkinson's disease (PD)
* At least 2 of 3 cardinal signs of PD
* Response to dopaminergic medication

Exclusion Criteria:

* Angina pectoris
* History of myocardial infarction within 6 months
* History of ventricular dysrhythmia requiring current therapy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David W Sparrow, DSc, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Structured Exercise | Lifestyle Exercise
Started | 89 | 80
Completed | 84 | 77
Not Completed | 5 | 3
Not completed — Death | 4 | 2
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Structured Exercise | Lifestyle Exercise | Total
Number analyzed (Participants) | 89 | 80 | 169
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.5 (9.4) | 72.7 (9.8) | 72.1 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 87 | 78 | 165
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Total Falls During the 1-year Follow-up
Description: Total number of falls over the 1-year follow-up; self-reported falls collected on a weekly basis and totaled over the follow-up period.
Time Frame: up to 1 year
Population: 2 participants not analyzed were excluded due to "early loss to follow-up" and had no fall data collected.
Measure: Number; unit: Total count of falls
Arm/Group | Structured Exercise | Lifestyle Exercise
Number analyzed (Participants) | 88 | 79
Total count of falls | 1026 | 1861
Statistical Analysis 1: Comparison: Structured Exercise vs Lifestyle Exercise; Testing to see if there is a significant difference in fall rates over 12months between the two groups; Test type: Superiority; p < 0.001, Negative Binomial Regression; Incidence Rate Ratio = 0.39, 95% CI 2-sided [0.22 to 0.68]

ADVERSE EVENTS:
Time Frame: Adverse events were collected over 1 year participation period.
Arm/Group | Structured Exercise | Lifestyle Exercise
All-Cause Mortality (participants affected / at risk) | 4/89 | 2/80
Serious Adverse Events (participants affected / at risk) | 4/89 | 2/80
Other Adverse Events (participants affected / at risk) | 0/89 | 0/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Structured Exercise (N=89) | Lifestyle Exercise (N=80)
Death (General disorders) | 4 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes